CLINICAL TRIAL: NCT06687083
Title: Non-Invasive High Frequency Oscillatory Ventilation Versus Continuous Positive Airway Pressure in Preterm Neonates with Respiratory Distress Syndrome
Brief Title: Nasal High Frequency in Preterm Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mariam Ibrahim, assistant professor of pediatrics, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: nasal high frequency neonates
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Respiratory Distress Syndrome (RDS); Neonatal Diseases and Abnormalities
Keywords: preterm neonate; non invasive ventilation; high frequency ventilation; respiratory distress
MeSH Terms: conditions — Respiratory Distress Syndrome; Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Dyspnea

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- nasal high frequency (Experimental): Preterm neonates who will be allocated will start nHFOV. nHFOV will be provided via binasal prongs (Size: small, medium, large; Diameter according to its chart.
  The initial parameters will be mean airway pressure (MAP) of 6 cm H2O (range 6-10), frequency of 8 Hz (range 8-12) and amplitude will be adjusted until infant's chest showed slight oscillations and amplitude will be 7 (range 7-10).
  The fraction of inspired oxygen (FiO2) will be adjusted to maintain target oxygen saturation (SpO2) from 92% to 95% by a pulse oximeter
  Interventions: Device: nasal high frequency oscillatory ventilation mode
- nasal CPAP (Active Comparator): Preterm neonates who will be allocated to this group to the nCPAP will be started on a pressure of 6-8 cm H2O, FiO2) will be adjusted to maintain target oxygen saturation (SpO2) from 92% to 95% by a pulse oximeter.
  Interventions: Drug: nasal continuous positive pressure ventilation mode

INTERVENTIONS:
Device: nasal high frequency oscillatory ventilation mode — Preterm neonates who will be allocated will start nHFOV: (CNO, Medin, Germany). nHFOV will be provided via binasal prongs (Size: small, medium, large; Diameter according to its chart; Medin, Germany).
  The initial parameters will be mean airway pressure (MAP) of 6 cm H2O (range 6-10), frequency of 8 Hz (range 8-12) and amplitude will be adjusted until infant's chest showed slight oscillations and amplitude will be 7 (range 7-10).
  The fraction of inspired oxygen (FiO2) will be adjusted to maintain target oxygen saturation (SpO2) from 92% to 95% by a pulse oximeter.
  Arms: nasal high frequency
Drug: nasal continuous positive pressure ventilation mode — Preterm neonates who will be allocated to this group to the nCPAP will be started on a pressure of 6-8 cm H2O, FiO2) will be adjusted to maintain target oxygen saturation (SpO2) from 92% to 95% by a pulse oximeter
  Arms: nasal CPAP

SUMMARY:
One of the most commonly used non-invasive methods is nasal continuous positive airway pressure (nCPAP). Although high frequency ventilation (HFV) has been applied in many neonatal intensive care units, nasal high frequency oscillatory ventilation (nHFOV) is a relatively new non-invasive modality. The application of nasal high-frequency ventilation with the strategy of lung recruitment will combine benefits of improving gas exchange and decreasing lung injury together with avoiding complication of invasive ventilation.

DETAILED DESCRIPTION:
Premature infants with respiratory distress syndrome (RDS) usually require respiratory support . Due to the complications of intubation and mechanical ventilation, in the last decade, attempts have been made to use non-invasive methods in the management of these patients . Over the past few decades, nasal ventilation has been used to control and improve respiratory failure in infants with RDS . nCPAP is a relatively simple and effective therapy in the early management of RDS in newborns . nCPAP is the application of positive pressure to the airways of spontaneously breathing neonates throughout the respiratory cycle . However, some neonates with this therapeutic approach also develop respiratory failure and need mechanical ventilatory support. According to some investigations, 43%-80% of infants with moderate to severe respiratory failure who are initially treated with nCPAP need mechanical ventilation .

In recent years, the beneficial effects of high-frequency ventilators (HFV) have been shown in the management of RDS as well as the use of this mode as the initial mode of support or as a rescue treatment after failure of conventional mechanical ventilation. In high-frequency ventilation, a low tidal volume with a higher frequency than that of physiological respiration is produced. This technique is very effective in eliminating carbon dioxide (CO2). Adequate recruitment of lung volume in this mechanical mode has the main role of protecting and preserving lung architecture as well as potentiating surfactant therapy.

The nHFOV is a non-invasive ventilation mode that applies an oscillatory pressure waveform to the airways using a nasal interface. nHFOV is effective and superior to nasal intermittent positive pressure ventilation in terms of lung CO2 elimination. This mode has been shown to facilitate CO2 elimination, but little is known about its use in neonates. There is increasing evidence of beneficial effects of nHFOV in reducing the duration of ventilator support compared with the effects of nCPAP in RDS. We intended to explore the benefits of nHFOV vs nCPAP in preterm neonates.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age: 30-34 weeks (determined by date of last menstrual period or ultrasound) and confirmed by Ballard score.
* Recruited immediately after birth Up to 24 hours of age.
* Appropriate weight for the gestational age.
* Spontaneous breathing and clinical signs and symptoms of respiratory distress syndrome (grunting, cyanosis, intercostal and subcostal retractions) or RDS Silverman Score > 5.

Exclusion Criteria:

* Major congenital abnormalities, congenital heart disease and diaphragmatic hernia.
* A need for intubation and mandatory ventilation during resuscitation or on the first day of life.
* Perinatal asphyxia (Umbilical cord pH < 7.16, and umbilical cord bicarbonate < 12 mEq/L)
* Pulmonary hemorrhage and severe intraventricular hemorrhage (IVH) on admission.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
need for invasive mechanical ventilation | five days

SECONDARY OUTCOMES:
duration of respiratory support | one month
mortality | one month

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
data can be shared upon accepted reasons
Supporting Information: Study Protocol

REFERENCES:
- [Background] Diblasi RM. Nasal continuous positive airway pressure (CPAP) for the respiratory care of the newborn infant. Respir Care. 2009 Sep;54(9):1209-35. PMID 19712498
- [Background] Aktas S, Unal S, Aksu M, Ozcan E, Ergenekon E, Turkyilmaz C, Hirfanoglu I, Atalay Y. Nasal HFOV with Binasal Cannula Appears Effective and Feasible in ELBW Newborns. J Trop Pediatr. 2016 Apr;62(2):165-8. doi: 10.1093/tropej/fmv088. Epub 2015 Dec 27. PMID 26710797